CLINICAL TRIAL: NCT07085390
Title: Balloon Guide Versus Conventional Guide Catheter in Stroke Thrombectomy
Acronym: 2Guide
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 007664
Record Dates: First submitted 2025-05-16; First posted 2025-07-25 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Acute Ischemic Stroke AIS
Keywords: Ischemic Stroke; Thrombectomy
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Balloon Guide Catheter (Other): Use of a balloon guide catheter in stroke thrombectomy.
  Interventions: Other: Use of a Balloon Guide Catheter
- Conventional Guide Catheter (Other): Use of conventional (non-balloon guide) catheter in stroke thrombectomy.
  Interventions: Other: Use of a Conventional (non-balloon) Guide Catheter

INTERVENTIONS:
Other: Use of a Balloon Guide Catheter — Use of a balloon guide catheter in stroke thrombectomy.
  Arms: Balloon Guide Catheter
Other: Use of a Conventional (non-balloon) Guide Catheter — Use of a conventional (non-balloon) guide catheter in stroke thrombectomy.
  Arms: Conventional Guide Catheter

SUMMARY:
The purpose of this clinical trial is to study the two main types of approaches used in stroke thrombectomy and to investigate if one approach is more effective than the other, as this is currently not known. This study will be conducted in adults who have been diagnosed with an acute ischemic stroke and who are undergoing a thrombectomy for the treatment of their stroke. The main questions it aims to answer are:

* Does the use of a balloon guide catheter versus a conventional guide catheter lower the time needed to restore blood flow in the blocked vessel in the brain
* To help researchers better understand the technical, clinical, and procedural outcomes associated with using a balloon guide catheter versus a conventional guide catheter in stroke thrombectomy

Participants will be asked to

* Share their medical history and imaging data that is collected as part of their routine medical care
* Undergo a mechanical thrombectomy as part of their routine medical care
* Answer some questions about their neurological functioning at 3 months (90 days) post hospitalization

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Patient is undergoing a stroke thrombectomy procedure at the enrolling hospital
* Patient or the legally authorized representative are able to provide signed informed cosent for the study
* Patient is not enrolled in another clinical trial that may interfere with the results or interpretation of this study
* Identification of a Large Vessel Occlusion (LVO) on imaging

Exclusion Criteria:

* Lack of signed informed consent from the patient or legally authorized representative
* Spontanous recanalization or any other reason in which the mechanical thrombectomy procedure would be terminated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
TICI Grading Scale Score | Participant duration is 90 days.
  Use of a mTICI grading scale to look at the degree to which the vessel has been opened during a mechanical thrombectomy.

SECONDARY OUTCOMES:
Procedural Outcomes | Participant duration is 90 days.
  Metrics associated with a standard of care thrombectomy procedure, such as length of procedure, will be collected.
Number of Participants with Treatment Related Adverse Effects | Participant duration is 90 days.
  Collection of data related to clincial and safety outcomes such as presence of a bleed.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Florida (USF), Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with participants as both catheters are routinely used in acute ischemic stroke thrombectomy. The decision to use a balloon guide versus a conventional guide catheter is usually left to the discretion of the operator.